CLINICAL TRIAL: NCT02350595
Title: Fiskespisestudiene 2011-2014. Spiseforsøk Med Fisk. Delstudie 2: Studie av Mulige Effekter av Fet og Mager Fisk på Glukosemetabolismen og inflammasjonsmarkører i Overvektige Voksne.
Brief Title: A Study on the Possible Health Effects of Lean Fish and Fatty Fish Intake in Overweight or Obese Adults
Acronym: FISK2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Bergen Medical Research Foundation (Other); Skretting ASA (Unknown); Leroy Seafood Group ASA (Industry)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Researcher, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FISK2
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — bearberry, bladderwrack, borage oil, centella, fatty acid, fish oil, ginkgo biloba, melilotus, soya lecithin drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lean fish (Experimental): Participants eat 750g of lean fish per week for 8 weeks.
  Interventions: Other: Lean fish
- Fatty fish (Experimental): Participants eat 750g of fatty fish per week for 8 weeks.
  Interventions: Other: Fatty fish
- Control (No Intervention): Participants eat as normal, but avoid fish and seafood for 8 weeks.

INTERVENTIONS:
Other: Lean fish
  Arms: Lean fish
Other: Fatty fish
  Arms: Fatty fish

SUMMARY:
The potential health effects of high intake of lean or fatty fish will be investigated in overweight or obese adults. Participants consume 750g/week of fillets of fish for 8 weeks.

Hypothesis:

High intake of fatty or lean fish will beneficially affect glucose regulation and the immune system.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥27 kg/m2
* fasting blood glucose ≤7.0 mmol/L

Exclusion Criteria:

* pregnancy
* incompatibility with fish consumption (allergies, intolerance and/or dislike)
* diagnosed diabetes mellitus, heart disease or gastrointestinal diseases
* use of medications affecting lipid metabolism or glucose homeostasis
* use of anti-inflammatory medications
* use of supplements containing long chain n-3 fatty acids
* intentional weight loss
* and large fluctuation in body weight (>3 kg) over the previous two months

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in serum concentrations of glucose | baseline and 8 weeks

SECONDARY OUTCOMES:
Changes in insulin, insulin C-peptide, leukocyte fatty acids, leukocyte function, body weight and composition, and intake of energy and macronutrients within the groups over time. | baseline and 8 weeks
Changes in serum vitamin concentrations after fish intake. | baseline and 8 weeks
  Serum concentrations of fat-soluble and water-soluble vitamins were measured, and dietary intakes of vitamins were estimated based on reported food intake from 5-day food diaries.
Changes in serum and urine concentrations of amino acids and metabolites of amino acids after fish intake. | baseline and 8 weeks
  Concentrations of amino acids and amino acid metabolites were measured in fasting serum and morning urine
Changes in fecal microbiota profile after fish intake. | baseline and 8 weeks
  54 DNA bacterial markers targeting more than 300 bacteria based on their 16S rRNA sequence in seven variable regions were analysed in feces (72h collection)
Changes in fecal and serum concentrations of lipids and bile acids after fish intake. | baseline and 8 weeks
  Fat, cholesterol and total bile acids were quantified in feces (72h collection) and fasting serum.
Changes in markers of oxidative stress after fish intake. | baseline and 8 weeks
  Antioxidant enzymes, antioxidant enzyme cofactors and biomarkers of oxidative stress were quantified in serum
Changes in total neopterin after fish intake | baseline and 8 weeks
  Total neopterin was measured in serum.
Quantification of markers of kidney dysfunction | baseline and 8 weeks
  Urine concentrations of cystatin C and T-cell immunoglobulin mucin-1 (relative to creatinine) were measured as markers of kidney function
Changes in amino acids and metabolites of amino acids after a standardized meal. | baseline
  Concentrations of amino acids and amino acid metabolites were measured in fasting and postprandial serum
Changes in metabolites and co-factors involved in one-carbon metabolism after a standardized meal | baseline
  Concentrations of relevant metabolites and co-factors were measured in fasting and postprandial serum
Comparisons of amino acid concentrations in serum and urine between men and women | baseline
  Concentrations of amino acids and amino acid metabolites were measured in serum and urine
Comparisons of metabolites and co-factors involved in one-carbon metabolism in serum and urine between men and women | baseline
  Concentrations of relevant metabolites and co-factors were measured in serum and urine

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Result] Helland A, Bratlie M, Hagen IV, Mjos SA, Sornes S, Ingvar Halstensen A, Brokstad KA, Sveier H, Rosenlund G, Mellgren G, Gudbrandsen OA. High intake of fatty fish, but not of lean fish, improved postprandial glucose regulation and increased the n-3 PUFA content in the leucocyte membrane in healthy overweight adults: a randomised trial. Br J Nutr. 2017 May;117(10):1368-1378. doi: 10.1017/S0007114517001234. Epub 2017 Jun 13. PMID 28606215
- [Result] Helland A, Bratlie M, Hagen IV, Midttun O, Sveier H, Mellgren G, Ueland PM, Gudbrandsen OA. Effect of high intake of cod or salmon on serum total neopterin concentration: a randomised clinical trial. Eur J Nutr. 2021 Sep;60(6):3237-3248. doi: 10.1007/s00394-021-02497-0. Epub 2021 Feb 12. PMID 33576844
- [Result] Bratlie M, Hagen IV, Helland A, Erchinger F, Midttun O, Ueland PM, Rosenlund G, Sveier H, Mellgren G, Hausken T, Gudbrandsen OA. Effects of high intake of cod or salmon on gut microbiota profile, faecal output and serum concentrations of lipids and bile acids in overweight adults: a randomised clinical trial. Eur J Nutr. 2021 Jun;60(4):2231-2248. doi: 10.1007/s00394-020-02417-8. Epub 2020 Oct 27. PMID 33108521
- [Result] Bratlie M, Hagen IV, Helland A, Midttun O, Ulvik A, Rosenlund G, Sveier H, Mellgren G, Ueland PM, Gudbrandsen OA. Five salmon dinners per week were not sufficient to prevent the reduction in serum vitamin D in autumn at 60 degrees north latitude: a randomised trial. Br J Nutr. 2020 Feb 28;123(4):419-427. doi: 10.1017/S0007114519002964. Epub 2019 Nov 25. PMID 31760958
- [Result] Hagen IV, Helland A, Bratlie M, Midttun O, McCann A, Sveier H, Rosenlund G, Mellgren G, Ueland PM, Gudbrandsen OA. TMAO, creatine and 1-methylhistidine in serum and urine are potential biomarkers of cod and salmon intake: a randomised clinical trial in adults with overweight or obesity. Eur J Nutr. 2020 Aug;59(5):2249-2259. doi: 10.1007/s00394-019-02076-4. Epub 2019 Aug 10. PMID 31401679
- [Derived] Hagen IV, Helland A, Bratlie M, Midttun O, McCann A, Ulvik A, Mellgren G, Ueland PM, Gudbrandsen OA. Serum concentrations of amino acids and tryptophan metabolites are affected by consumption of a light breakfast: a clinical intervention study in adults with overweight or obesity. BMC Nutr. 2023 Jan 11;9(1):10. doi: 10.1186/s40795-022-00661-1. PMID 36631895